CLINICAL TRIAL: NCT07353385
Title: Enhanced Efficacy Through Optimization of Hemoporfin-Photodynamic Therapy Parameters in Port-Wine Stains: A Prospective, Randomized Controlled Study
Brief Title: Enhanced Efficacy Through Optimization of Hemoporfin-Photodynamic Therapy Parameters in Port-Wine Stains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Weihui Zeng, Professor, Second Affiliated Hospital of Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024219
Record Dates: First submitted 2025-12-30; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Port Wine Stains
MeSH Terms: conditions — Hemangioma, Capillary

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low power group (Experimental): Received irradiation at 75 mW/cm² for 19 minutes per spot.
  Interventions: Radiation: irradiation at 75 mW/cm² for 19 minutes per spot
- High power group (Experimental): Received irradiation at 84 mW/cm² for 17 minutes per spot.
  Interventions: Radiation: irradiation at 84 mW/cm² for 17 minutes per spot

INTERVENTIONS:
Radiation: irradiation at 84 mW/cm² for 17 minutes per spot — Patients were positioned appropriately, with pediatric patients secured using a restraining bed. The target lesions were fully exposed (shaved if necessary), cleansed, disinfected, and the surrounding healthy skin was shielded with black cloth. The laser parameters and handpiece position were adjusted to ensure the lesion remained within the effective irradiation field.
  Under dim light, a prepared Hemoporfin (Shanghai Fudan Zhangjiang Pharmaceutical Co., Ltd.) solution was diluted to 20 mL at a dosage of 5.0 mg/kg and administered via infusion pump at a controlled rate within 5 minutes. Approximately 3 minutes post-initiation of infusion, irradiation with a 532-nm LED green light (Wuhan Yage Optoelectronic Technology Co., Ltd.) commenced. To maintain an identical total light dose between groups, the high-power group received 84 mW/cm² for 17 minutes per spot.
  Arms: High power group
Radiation: irradiation at 75 mW/cm² for 19 minutes per spot — Patients were positioned appropriately, with pediatric patients secured using a restraining bed. The target lesions were fully exposed (shaved if necessary), cleansed, disinfected, and the surrounding healthy skin was shielded with black cloth. The laser parameters and handpiece position were adjusted to ensure the lesion remained within the effective irradiation field.
  Under dim light, a prepared Hemoporfin (Shanghai Fudan Zhangjiang Pharmaceutical Co., Ltd.) solution was diluted to 20 mL at a dosage of 5.0 mg/kg and administered via infusion pump at a controlled rate within 5 minutes. Approximately 3 minutes post-initiation of infusion, irradiation with a 532-nm LED green light (Wuhan Yage Optoelectronic Technology Co., Ltd.) commenced. To maintain an identical total light dose between groups, the low-power group received 75 mW/cm² for 19 minutes per spot.
  Arms: Low power group

SUMMARY:
1. Background and Objectives Port-wine stain (PWS) is a congenital capillary malformation located in the upper dermis. Hematoporphyrin monomethyl ether (HMME)-mediated photodynamic therapy (PDT) has been established as a primary and effective treatment for PWS in China. However, treatment parameters, particularly irradiance and irradiation duration, vary widely in clinical practice based on physician experience, with a lack of evidence from controlled trials to guide optimization. The efficacy of PDT relies on a type II photochemical reaction, which is oxygen-dependent. High irradiance may lead to rapid oxygen depletion in the treatment area, potentially limiting therapeutic outcomes. This prospective, randomized controlled trial aims to compare the efficacy and safety of a low-irradiance, prolonged-duration protocol versus a high-irradiance, shorter-duration protocol in HMME-PDT for PWS, while maintaining an identical total light dose.
2. Study Design

   This was a single-center, randomized controlled, single-blind trial. The study protocol was approved by the Ethics Committee of The Second Affiliated Hospital of Xi'an Jiaotong University (Approval No. 2024219). A total of 33 pediatric patients (aged 3-12 years) with facial or neck PWS were enrolled and randomly assigned to one of two groups:

   Low-Power Group (n=15): Received irradiation at 75 mW/cm² for 19 minutes per spot.

   High-Power Group (n=18): Received irradiation at 84 mW/cm² for 17 minutes per spot.

   Both groups received a single session of HMME-PDT with the same total light dose. All patients received an intravenous infusion of Hemoporfin at a dose of 5.0 mg/kg, followed by irradiation with a 532-nm LED green light.
3. Primary evaluation indicators

The primary efficacy endpoint was lesion clearance assessed at the 3-month follow-up using three independent methods:

Blinded Quartile Grading: Performed by two independent dermatologists based on high-resolution photographs.

Quantitative Lesion Area Reduction: The percentage reduction in the PWS area was calculated from VISIA complexion analysis system "redness" images using ImageJ software.

Erythema Index (EI) Analysis: The relative change in the EI (ΔEI%) between the lesion and normal skin was quantified.

ELIGIBILITY:
Inclusion Criteria:

·Clinical diagnosis of port-wine stain (PWS).

Exclusion Criteria:

* concurrent syndromes such as Sturge-Weber or Klippel-Trenaunay syndrome;
* a history of previous radiotherapy, photodynamic therapy, or any other intervention in the treatment area that might confound efficacy evaluation;
* a known diagnosis of cutaneous photosensitivity, porphyria, or hypersensitivity to porphyrin-based drugs;
* administration of photosensitizing medications, including but not limited to griseofulvin, retinoids, thiazide diuretics, sulfonamides, and tetracyclines, within 4 weeks prior to the study.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Blinded Quartile Grading | from enrollment to 3 months post-treatment
  Clinical efficacy was assessed by two blinded dermatologists using a quartile grading scale based on high-resolution photographs taken before treatment and at the 3-month follow-up. Therapeutic responses were classified into four grades: an Excellent Response was defined as lesion clearance of 75% or greater; a Good Response represented clearance ranging from 50% to 74%; a Moderate Response indicated clearance between 25% and 49%; and a Poor Response was assigned for clearance of 24% or less.

SECONDARY OUTCOMES:
Quantitative Lesion Area Reduction | from enrollment to 3 months post-treatment
  Objective evaluation was performed by analyzing the VISIA-captured "redness images" with ImageJ software (National Institutes of Health), where the percentage reduction in the lesion area was calculated.
Erythema Index (EI) Analysis | from enrollment to 3 months post-treatment
  The relative change in the EI (ΔEI%) between the lesion and normal skin was quantified. The standardized VISIA images were imported into ImageJ and split into RGB channels. The R (red) and G (green) channels were subsequently converted into logarithmic images. An 'EI image' was generated by subtracting the Log G image from the Log R image using the Image Calculator function. The mean EI values were then measured within both the lesion and an adjacent normal skin area. The differences (ΔEI) were calculated as follows: ΔEIpre = EIlesion(pre) - EInormal(pre); ΔEIpost = EIlesion(post) - EInormal(post). The final improvement percentage was expressed as ΔEI% = (ΔEIpre - ΔEIpost) / ΔEIpre × 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Xi'an Jiao Tong University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided